CLINICAL TRIAL: NCT03533907
Title: Pregnancy Outcomes in Infertile Patients After Treatment With Ulipristal Acetate: Preliminary Academic Assisted Reproductive Technology Center Experience.
Brief Title: Pregnancy Outcomes in Infertile Patients After Treatment With Ulipristal Acetate.
Status: Completed | Type: Observational
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Sponsor
Other Study IDs: 8/2018
Record Dates: First submitted 2018-05-11; First posted 2018-05-23 (Actual); Last update posted 2018-06-08 (Actual); Status verified 2018-05

CONDITIONS: Myoma;Uterus; Infertility, Female
MeSH Terms: conditions — Myofibroma; Infertility, Female

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- treated: The women included were patients of the Humanitas Fertility Center; they all had a diagnosis of infertility and were trying to become pregnant. They received ≥1 month of therapy with UA 5 mg/day

SUMMARY:
The investigators analyzed a group of infertile women treated with Ulipristal Acetate (UA) for uterine fibroids at the Humanitas Fertility Center. All the patients' data were extracted from the Fertility Center external-audit-anonymized electronic research query system.

DETAILED DESCRIPTION:
In the recent years several large studies have been published on the efficacy of Ulipristal Acetate treatment of moderate to severe symptoms of uterine fibroids in adult women: initially proposed only as pre-surgical treatment, the UA was subsequently also used for the long-term treatment of uterine myomas symptoms.

However, few data are available on the effects of UA in terms of increasing fecundability, implantation and pregnancy outcome and safety in the general population, and in infertile patients in particular.

This retrospective study aims at describing the correlation between the use of Ulipristal Acetate and pregnancy outcome in infertile patients and at comparing the UA plus surgery approach to the UA-only treatment in terms of pregnancy outcome.

ELIGIBILITY:
Inclusion Criteria:

* infertile women received at least 1 month of therapy with UA 5 mg/day for uterine fibroids
* more of 1 year of active pregnancy seeking

Exclusion:

* menopausal women;

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Study Population: The women included were patients of the Humanitas Fertility Center; they all had a diagnosis of infertility and were trying to become pregnant. They received ≥1 month of therapy with UA 5 mg/day over the period 2013 - 2018
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2013-11-01 (Actual); Primary Completion 2018-04-10 (Actual); Study Completion 2018-05-01 (Actual)

PRIMARY OUTCOMES:
implantation rate | 2013 - 2018
  number of intrauterine gestational sacs observed divided by the number of transferred embryos

SECONDARY OUTCOMES:
myomas reduction | 2013 - 2018
  volumetric reduction in after therapy

CONTACTS AND LOCATIONS:
Locations (1):
- Paolo Emanuele Levi Setti, Rozzano, MI, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Luyckx M, Squifflet JL, Jadoul P, Votino R, Dolmans MM, Donnez J. First series of 18 pregnancies after ulipristal acetate treatment for uterine fibroids. Fertil Steril. 2014 Nov;102(5):1404-9. doi: 10.1016/j.fertnstert.2014.07.1253. Epub 2014 Sep 17. PMID 25241376
- [Result] Donnez J, Donnez O, Matule D, Ahrendt HJ, Hudecek R, Zatik J, Kasilovskiene Z, Dumitrascu MC, Fernandez H, Barlow DH, Bouchard P, Fauser BC, Bestel E, Loumaye E. Long-term medical management of uterine fibroids with ulipristal acetate. Fertil Steril. 2016 Jan;105(1):165-173.e4. doi: 10.1016/j.fertnstert.2015.09.032. Epub 2015 Oct 23. PMID 26477496